CLINICAL TRIAL: NCT06511609
Title: Comparison of Anti-reflux Effects of Laparoscopic Proximal Gastrectomy With Double-flap Technique (Kamikawa Anastomosis) Versus Double-tract Reconstruction: A Prospective, Multicenter, Randomized Controlled Trial.
Brief Title: The Anti-reflux Effect of Double-flap Technique in Laparoscopic Proximal Gastrectomy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhi People's Hospital Affiliated to Changzhi Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZPH-0001
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-05

CONDITIONS: Proximal Early Gastric Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double-flap technique（DFT） (Experimental): Laparoscopic proximal gastrectomy with double flap anastomosis group
  Interventions: Procedure: double-flap technique（DFT）; double-tract reconstruction(DTR),
- double-tract reconstruction（DTR） (Active Comparator): Laparoscopic proximal gastrectomy with double-tract anastomosis group
  Interventions: Procedure: double-flap technique（DFT）; double-tract reconstruction(DTR),

INTERVENTIONS:
Procedure: double-flap technique（DFT）; double-tract reconstruction(DTR), — DFT (experiment group). Patients receive double flap technique after laparoscopic proximal gastrectomy. DTR (control group). Patients receive double-tract reconstruction after laparoscopic proximal gastrectomy.

SUMMARY:
This study is a multicenter, open-label, prospective, randomized parallel-controlled trial. The purpose is to explore whether the incidence rate of reflux esophagitis (RE) within 12 months after surgery is non-inferior for the DFT group compared to the DTR group.

DETAILED DESCRIPTION:
This study will enroll patients with proximal gastric cancer scheduled to undergo laparoscopic proximal gastrectomy. The patients will be randomly divided into two groups. One group will undergo laparoscopic proximal gastrectomy with double-flap technique (DFT) anastomosis, while the other group will undergo laparoscopic proximal gastrectomy with double-tract reconstruction (DTR). The primary endpoint is the proportion of patients who develop reflux esophagitis within 12 months after surgery. The secondary endpoints include postoperative complications, surgery-related indicators, and postoperative nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 80 years, regardless of gender;
2. Patients diagnosed with gastric cancer through tissue biopsy;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
4. American Society of Anesthesiologists (ASA) classification of I to III;
5. Acceptable for laparoscopic proximal gastrectomy with preoperative examinations (based on endoscopic ultrasound and/or contrast-enhanced computed tomography of the thorax and abdomen) confirming the following oncological features:

   Primary tumor located in the upper part of the stomach (proximal 1/3 of the stomach) or gastroesophageal junction; Length of esophageal invasion ≤ 1 cm, tumor maximum diameter ≤ 4 cm; Preoperative staging T1-3N0M0 (based on AJCC 8th edition TNM clinical staging);
6. Voluntary signing of informed consent.

Exclusion Criteria:

1. Received preoperative chemotherapy, radiotherapy, targeted therapy, or immunotherapy;
2. Presence of contraindications to surgery;
3. Multiple malignant lesions in the stomach;
4. Presence of other malignancies that may affect the preservation of stomach function;
5. Previous upper abdominal surgery (excluding cholecystectomy);
6. Preoperative examination reveals active peptic ulcer;
7. Patients who have received or are currently receiving treatment for systemic inflammatory diseases;
8. Pregnant or breastfeeding women;
9. Conditions deemed unsuitable for participation in this study by the investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with reflux esophagitis | Within 12 months after surgery
  The percentage (%) of patients developing postoperative reflux esophagitis after surgery in the two group.

SECONDARY OUTCOMES:
Postoperative complications | Within 12 months after surgery
  Evaluated using the Clavien-Dindo classification to assess the severity of postoperative complications.
Operation time | Perioperative period
  From the beginning of surgery to the end of surgery
Kamikawa anastomosis time | Perioperative period
  The time of making the seromuscular flap and the time of esophagogastrostomy were included
intraoperative blood loss | Perioperative period
  The operation begins to end the amount of bleeding.
Weight change | Within 12 months after surgery
  Calculated in kilograms
Body Mass Index (BMI) | Within 12 months after surgery
  weight and height will be combined to report BMI in kg/m^2
Albumin value | Within 12 months after surgery
  The concentration of albumin in the blood, expressed in g/L.
Pre albumin value | Within 12 months after surgery
  The concentration of pre albumin in the blood, expressed in g/L.
Hemoglobin value | Within 12 months after surgery
  The concentration of Hemoglobin in the blood, expressed in g/L.
Folic acid value | Within 12 months after surgery
  The concentration of Folic acid value in the blood, expressed in ng/mL.
Vitamin B12 value | Within 12 months after surgery
  The concentration of Vitamin B12 value in the blood, expressed in uug/L.
Ferritin value | Within 12 months after surgery
  The concentration of Vitamin B12 value in the blood, expressed in ug/L.
Nutritional risk screening 2002 | Within 12 months after surgery
  The nutritional status is assessed using the Nutrition Risk Screening 2002 (NRS-2002) scale, with a scoring range of 0 to 7 points. A higher score indicates a worse nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: WenQing Hu, Study Chair — 502 Changxing Middle Road, Luzhou District, Changzhi City, Shanxi Province, China